CLINICAL TRIAL: NCT04350502
Title: Pharmacokinetics and Pleural Fluid Penetration of Amoxicillin and Clavulanic Acid in Patients With Pleural Infections
Acronym: PK-plèvre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0002
Record Dates: First submitted 2020-04-09; First posted 2020-04-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Pleural Infection; Empyema; Community-acquired Pneumonia; Pharmacokinetic; Amoxicillin
Keywords: Pleural Infection; Empyema; Community-acquired Pneumonia; pharmacokinetic; amoxicillin; clavulanic acid; pneumococcal antigen
MeSH Terms: conditions — Empyema; Community-Acquired Pneumonia | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- complicated pleural infection patients (Experimental): Patients with a complicated pleural infection will be managed according to the French guideline with a chest tube drainage associated to a treatment with amoxicillin (2g*3 by day) and clavulanic acid (200mg*3 by day). Repeated samples of pleural fluid and serum will be taken to evaluate antibiotics' concentrations at H0; H½; H1; H2; H3; H4; H8 and H24
  Interventions: Procedure: chest tube drainage; Biological: antibiotic concentration in pleural fluid; Drug: Amoxicillin + clavulanic acid

INTERVENTIONS:
Procedure: chest tube drainage — Patients with a complicated pleural infection will be managed according to the French guideline with a chest tube drainage associated to a treatment with amoxicillin (2g*3 by day) and clavulanic acid (200mg*3 by day).
Biological: antibiotic concentration in pleural fluid — Patients with a complicated pleural infection will be managed according to the French guideline with a chest tube drainage associated to a treatment with amoxicillin (2g*3 by day) and clavulanic acid (200mg*3 by day). Repeated samples of pleural fluid and serum will be taken to evaluate antibiotics' concentrations at H0; H½; H1; H2; H3; H4; H8 and H24
Drug: Amoxicillin + clavulanic acid — Patients with a complicated pleural infection will be managed according to the French guideline with a chest tube drainage associated to a treatment with amoxicillin (2g*3 by day) and clavulanic acid (200mg*3 by day). Repeated samples of pleural fluid and serum will be taken to evaluate antibiotics' concentrations at H0; H½; H1; H2; H3; H4; H8 and H24

SUMMARY:
The incidence of pleural infection is increasing worldwide since the last two decades. Antibiotics are one of the cornerstones of the treatment of this disease and must be associated to a correct evacuation of the pleural effusion.

Data concerning the pleural diffusion of antibiotics currently used in community acquired pleural infection are scarce. The main objective of this study is to evaluate the pleural pharmacokinetic of amoxicillin and clavulanic acid in patients with a complicated pleural infection (patients who need a chest tube insertion).

DETAILED DESCRIPTION:
Only scarce data are known on the pleural diffusion of antibiotics. Most of these data are concerning antibiotics that are not commonly used for the treatment of community-acquired pleural infections. Moreover, these data are obtained from studies using heterogenous methodologies (single or repeated evaluation of the antibiotic concentration in the pleural effusion, with or without correlation to the serum concentration; animal model or very specific population (i.e. uninfected patients or following lung surgery).

The main objective of this study is to evaluate the pleural pharmacokinetic of amoxicillin and clavulanic acid in patients with a community-acquired complicated pleural infection.

Patients with a complicated pleural infection will be managed according to the French guideline with a chest tube drainage associated to a treatment with amoxicillin (2g*3 by day) and clavulanic acid (200mg*3 by day). Repeated samples of pleural fluid and serum will be taken to evaluate antibiotics' concentrations at H0; H½; H1; H2; H3; H4; H8 and H24.

The follow-up and management of the included patients will not be modified by the study protocol except for the pleural and serum samples. Clinical, biological and radiological (chest x-ray and/or thoracic ultrasound) evaluation will be performed daily. Success of the pleural drainage will be assessed at day 3.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients (≥ 18 years old) hospitalized for a complicated community acquired pleural infection at University Hospital Amiens-Picardie.
* Complicated pleural infection is defined by the presence of one of the following criteria: frank pus, loculated pleural fluid, presence of organisms identified by Gram stain and/or culture from a non-purulent pleural fluid sample, pleural fluid pH <7.2, pleural fluid glucose <0.32g/l or large non-purulent effusion.

Exclusion Criteria:

* non-infectious pleural effusion
* hospital-acquired pleural infection
* patient treated with amoxicillin and clavulanic acid (if treatment was started more than > 24h ago)
* Minors, pregnant women, adult patients protected by law.
* Pleural infection requiring instant thoracic surgery
* allergy to beta-lactam
* Injection of contrast agent (Iomeron or Iohexol) during the 24 hours preceding or following the first dose of amoxicillin / clavulanic acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Pleural Concentration Versus Time Curve (AUC) of "amoxicillin and clavulanic acid" | up to 72 hours after starting chest pleural drainage
  Area Under the Pleural Concentration Versus Time Curve (AUC) of "amoxicillin and clavulanic acid" in patients with a complicated pleural infection

CONTACTS AND LOCATIONS:
Overall Officials: Damien BASILLE, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No